CLINICAL TRIAL: NCT01173978
Title: Insulinotropic Effect of GIP and GLP-1 Before and After Reduced Glucose Induced by Steroid Treatment, Relative Physical Inactivity and High Calorie Diet
Brief Title: Insulinotropic Effect of GIP and GLP-1 Before and After Reduced Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); European Foundation for the Study of Diabetes (Other)
Responsible Party: Katrine Bagge Hansen. MD, Glostrup University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: DYS-CLAMP
Record Dates: First submitted 2010-06-07; First posted 2010-08-03 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2010-07

CONDITIONS: Insulin Resistance; Deteriorated Glucose Homeostasis; Inactivity
Keywords: Incretin hormones; Glucagon; Insulin/c-peptide; Plasma glucose; Insulin resistance; Deteriorated glucose homeostasis; Inactivity
MeSH Terms: conditions — Insulin Resistance; Sedentary Behavior | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (Experimental): Each participant is examined during a normal, active lifestyle, without any intervention: The examinations include an OGTT, a glucagon test, three hyperglycemic clamps with infusion of a)GLP-1; b)GIP; c)Nacl
  Interventions: Other: No intervention
- Intervention (Experimental): Each participant is examined during a 12 days intervention.The examinations include an OGTT, a glucagon test, three hyperglycemic clamps with infusion of a)GLP-1; b)GIP; c)Nacl
  Interventions: Behavioral: Steroid hormone

INTERVENTIONS:
Behavioral: Steroid hormone — Steroid hormone: 37,5 mg of prednisolone; High energy diet: 130 % of recommended daily energy intake; Relative physical inactivity: no exercise and at least 8 hours of rest/day
  Other Names: Prednisolone
  Arms: Intervention
Other: No intervention
  Arms: No intervention

SUMMARY:
The incretin effect in patients with type two diabetes is reduced. The investigators have previously shown that it is possible to induce a defect in the incretin effect in healthy individuals. The purpose of this study is to evaluate the insulinotropic affect of the incretin hormones in healthy individuals before and after a deterioration of the glucose homeostasis.

DETAILED DESCRIPTION:
The incretin effect in patients with type two diabetes is reduced. The investigators have previously shown that it is possible to induce a defect in the incretin effect in healthy individuals. The purpose of this study is to evaluate the insulinotropic affect of the incretin hormones in healthy individuals before and after a deterioration of the glucose homeostasis. The evaluation is done by infusing GIP, GLP-1 or saline during hyperglycemic clamps.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians without type 2 diabetes mellitus
* Normal OGTT (75 g of glucose) according to WHO's criteria
* BMI 20-30
* Hemoglobin > 8.0 mmol/l
* Informed consent

Exclusion Criteria:

* Liver disease (ALAT > 2 x normal level)
* Nephropathy (s-creatinin > 130 µM or albuminuria)
* Relatives (parents/siblings) with T2DM
* Medical treatment witch cannot be stopped for 12 hours

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Insulinotropic effect of incretin hormones | 12 days
  Measurements of the insulinotropic effect of incretin hormones before and after 12 days intervention with steroid treatment, high calorie diet and relative physical inactivity

SECONDARY OUTCOMES:
Plasma concentration of glucagon | 12 days
  Measurements of plasma concentration of glucagon before and after 12 days intervention with steroid treatment, high calorie diet and relative physical inactivity

CONTACTS AND LOCATIONS:
Overall Officials: Katrine B Hansen, MD, Principal Investigator — Glostrup University Hospital; Filip K Knop, MD,PhD, Study Chair — Gentofte University Hospital; Tina Vilsbøll, MD,DmSc, Study Chair — Gentofte University Hospital; Jens J Holst, MD, DmSc, Study Chair — University of Copenhagen
Locations (1):
- Department of Clinical Physiology, Glostrup Municipality, Denmark